CLINICAL TRIAL: NCT06181032
Title: A Single-arm Prospective Clinical Study of Adebrelimab in Combination With Apatinib Gemcitabine and Cisplatin for the Neoadjuvant Treatment of Biliary Tract Malignancies
Brief Title: A Study of Adebrelimab in Combination With Apatinib Gemcitabine and Cisplatin in Biliary Tract Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Zhang Zhibo, Director of Hepatobiliary and Pancreatic Surgery Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-FJ-BTC-II-001
Record Dates: First submitted 2023-11-23; First posted 2023-12-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Biliary Tract Malignancies
Keywords: biliary tract malignancies; neoadjuvant treatment; adebrelimab; apatinib; gemcitabine and cisplatin
MeSH Terms: interventions — apatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Neoadjuvant treatment with adebrelimab in combination with apatinib gemcitabine and cisplatin
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab: 1200mg or 20mg/kg, iv, D1, Q3W;
  Other Names: SHR-1316
Drug: Apatinib — Apatinib: 250 mg, po, QD, Q3W;
Drug: Gemcitabine — Gemcitabine: 1000 mg/m2, iv, 30min, D1, D8, Q3W;
Drug: Cisplatin — Cisplatin: 25 mg/m2, iv, 30min, D1, D8, Q3W; Injection sequence: adebelizumab → gemcitabine → cisplatin (sequential interval of at least 30 min), 3 cycles of neoadjuvant therapy.

SUMMARY:
Evaluating the efficacy and safety of adebrelimab in combination with apatinib, gemcitabine and cisplatin in the neoadjuvant treatment of patients with biliary tract malignancies.

DETAILED DESCRIPTION:
Existing immune-combination chemotherapy has shown excellent data in advanced biliary malignancies, so what is the efficacy and safety of this regimen in neoadjuvant therapy? Moreover, the current combination model of immunization combined with anti-angiogenic drugs has become another new direction in the field of solid tumor treatment. Therefore, our group designed a single-arm, prospective clinical study of adebrelimab in combination with apatinib, gemcitabine and cisplatin in the neoadjuvant treatment of biliary malignancies, aiming at evaluating the efficacy and safety of adebrelimab in combination with apatinib, gemcitabine and cisplatin in the neoadjuvant treatment of biliary malignancies in patients with a view to bringing longer-term benefits to patients with resectable biliary malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 years old ≤ 75 years old, both male and female.
* 2. Patients with gallbladder cancer or cholangiocarcinoma (intrahepatic or extrahepatic) diagnosed by histologic or cytologic examination.
* 3. high-quality cross-sectional imaging by computed tomography (CT) or magnetic resonance imaging (MRI) with a diagnosis of surgically resectable high-risk biliary malignancy limited to the liver, bile ducts, and/or regional lymph nodes. (Must meet at least one of the following criteria)
* (1) T-grade ≥ Ib (Ib-IV);
* (2) Single lesion > 5 cm;
* (3) Multifocal tumors or satellite lesions confined to the same hepatic lobe as the primary lesion but still technically resectable;
* (4) Presence of major vascular invasion but still technically resectable;
* (5) Suspected or involved regional lymph nodes (N1);
* (6) No distant extrahepatic disease (M0).
* 4. Patients who have not received previous systemic therapy and who, in the judgment of the physician, have no contraindications to surgery, and the patient agrees to undergo radical surgical treatment.
* 5. At least one measurable lesion (according to the RECIST 1.1 criteria requires that the measurable lesion be ≥10 mm in long diameter on spiral CT scan or ≥15 mm in short diameter in malignant lymph nodes).
* 6. ECOG PS score of 0-1.
* 7. Expected survival ≥ 12 weeks.
* 8. Normal function of major organs and fulfillment of the following criteria:
* (1) Criteria for routine blood tests need to be met: (no blood transfusion within 14 days)
* a. Hemoglobin (HB) ≥ 90g/L;
* b. White blood cell count (WBC) ≥3×109/L;
* c. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
* d. Platelet (PLT) ≥80×109/L.
* (2) Biochemical tests need to meet the following criteria:
* a. Bilirubin (BIL) <1.5 times the upper limit of normal (ULN);
* b. Glutamine aminotransferase (ALT) and glutamine aminotransferase AST <5 ULN;
* c. serum creatinine (Cr) ≤ 1.5 ULN.
* 9. Women of childbearing potential must have a negative pregnancy test (serum) or urine HCG test within 7 days prior to enrollment and be willing to use an appropriate method of contraception for the duration of the trial and for 8 weeks after the last administration of the test drug; in the case of males, they should be surgically sterilized or agree to use an appropriate method of contraception for the duration of the trial and for 8 weeks after the last administration of the test drug.
* 10. Subjects voluntarily enroll in the study, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria:

* 1. Pregnant or lactating women.
* 2. Patients with autoimmune diseases, organ/hematopoietic stem cell transplantation or other malignant tumors (except cured basal cell carcinoma of the skin and cervical carcinoma in situ).
* 3. Patients with impaired consciousness or inability to cooperate with treatment, or patients with combined mental illness.
* 4. Patients who have participated in other clinical trials in the last three months.
* 5. Patients who have received other PD-1, PD-L1, CTLA-4 inhibitors in the past.
* 6. Patients who have undergone major surgery or chemotherapy or other systemic or localized treatments (including but not limited to radiation therapy, ablation therapy, etc.) for the target lesion prior to enrollment.
* 7. Use of interferon or systemic hormone therapy for immunosuppression within 14 days prior to enrollment (dose >10mg/day prednisone or other equipotent hormone).
* 8. Prior hypersensitivity to PD-1, PD-L1, CTLA-4 monoclonal antibody, any component of a chemotherapeutic agent, or other drugs of the same type used in the trial.
* 9. Bleeding from ruptured esophageal (fundus) varices within 1 month prior to treatment.
* 10. Uncorrectable coagulation dysfunction and serious blood abnormalities with severe bleeding tendency. Platelet count <50×109/L and severe coagulation abnormality cannot withstand surgery (anticoagulation therapy and/or anticoagulant application should be discontinued for more than 1 week before radiation therapy).
* 11. Intractable large amount of ascites and pleural fluid, malaise.
* 12. Severe liver, kidney, heart, lung, brain and other major organ failure.
* 13. Suffer from high blood pressure which cannot be reduced to normal range by antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg).
* 14. Previous severe cardiovascular disease, including but not limited to the following: myocardial ischemia or myocardial infarction of grade II or above, poorly controlled arrhythmia (including QTc interval ≥450 ms for men and ≥470 ms for women); cardiac insufficiency of grades Ⅲ to Ⅳ according to the NYHA standard or cardiac ultrasound suggesting that the left ventricular ejection fraction (LVEF) is <50%.
* 15. Patients with positive urine protein (urine protein test of 2+ or more, or 24-hour urine protein quantification >1.0g).
* 16. Inability to swallow tablets, malabsorption syndrome, or any condition that interferes with gastrointestinal absorption.
* 17. Patients with other serious concomitant conditions that, in the judgment of the investigator, jeopardize patient safety or interfere with the patient's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2029-02-23 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival（RFS） | 3 years
  Means the time from the date of the curative surgery to the date of relapse or death.
AE | 3 years
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

SECONDARY OUTCOMES:
Pathological complete response rate (pCR) | Within one week after surgery
  Rate of residual tumor cells not detected by pathology in excised tissue samples.
Major pathological response rate (MPR) | Within one week after surgery
  The percentage of active tumor cells in excised tissue samples is less than 10% of the rate.
surgery rate | Within one week after surgery
  Proportion of patients with final surgical resection among enrolled surgically resectable patients.
Radical (R0) resection rate | Within one week after surgery
  No residual cancer cells on the margins
Objective response rate (ORR) | Within 2 weeks prior to surgery
  Refers to the proportion of all subjects with a best overall result (BOR) of complete remission (CR) or partial remission (PR) as rated according to RECIST 1.1 criteria. If efficacy of CR or PR is achieved, subjects must be confirmed not less than 4 weeks ± 7 days after the initial evaluation.
Disease control rate (DCR) | Within 2 weeks prior to surgery
  Refers to the proportion of all subjects with a best overall result (BOR) of complete remission (CR), partial remission (PR), and stable disease (SD) as rated according to RECIST 1.1 criteria.
Overall survival (OS) | 5 years
  Defined as the time between the date of first dose and the death of the subject due to all causes. Subjects who were alive at the last follow-up visit had OS counted as data censored at the time of the last follow-up visit. The OS of subjects who were lost to follow-up was counted as data censored at the time of last confirmed survival prior to the lost follow-up. OS for data censoring was defined as the time from first dose to censoring.

CONTACTS AND LOCATIONS:
Overall Officials: Yufeng Chen, Principal Investigator — Zhangzhou Hospital of Fujian Medical University; Maolin Yan, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No